CLINICAL TRIAL: NCT06330792
Title: Effect of Bio-mechanical Awareness and Core Stability Exercises on Mechanical Low Back Pain Among Egyptian Physiotherapists
Brief Title: Effect of Bio-mechanical Awareness and Core Stability Exercises on Mechanical Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahim Ahmed Baza, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mechanical low back pain
Record Dates: First submitted 2024-03-13; First posted 2024-03-26 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Mechanical Low Back Pain
Keywords: mechanical awareness; core stability exercises
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Physiotherapists will be randomly subdivided into two equal groups in number. Group (A) (Experimental Group): This group will receive biomechanical awareness advices while working and core stability exercises.
  Group (B) (Control Group): This group will receive core stability exercises only.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effect of biomechanical awareness and core stability exercises on mechanical low back pain (Other)
  Interventions: Other: bio-mechanical awareness; Other: core stability exercises
- effect core stability exercises on mechanical low back pain (Other)
  Interventions: Other: core stability exercises

INTERVENTIONS:
Other: bio-mechanical awareness — Biomechanical awareness advices for physiotherapists during session: consist of group of awareness advices and McKenzie extension part method exercises to help physiotherapist working in correct position and consume his energy.
  Arms: effect of biomechanical awareness and core stability exercises on mechanical low back pain
Other: core stability exercises — Core stabilization exercise Program: The procedure for core stabilization exercises to improve core muscles in lumbar area

SUMMARY:
investigate the effect of bio-mechanical awareness and core stability exercises on mechanical low back pain among Egyptian Physiotherapists

DETAILED DESCRIPTION:
The aims of this study are:

1. to investigate the effect of bio-mechanical awareness and core stability exercises on the intensity of low back pain among Egyptian Physiotherapists.
2. to investigate the effect of bio-mechanical awareness and core stability exercises on and back muscle endurance among Egyptian Physiotherapists.
3. to investigate the effect of bio-mechanical awareness and core stability exercises on level of function (disability) associated with low back pain among Egyptian Physiotherapists.
4. to investigate the effect of bio-mechanical awareness and core stability exercises on fatigue among Egyptian Physiotherapists.
5. to investigate the effect of bio-mechanical awareness and core stability exercises on psycho-social factors at work among Egyptian Physiotherapists.

ELIGIBILITY:
inclusion criteria:

* Egyptian Physiotherapists with non-specific low back pain.
* Physiotherapy graduate who worked for at least two years (Khairy et al.,2019).
* Age range from 25 to 40 years old (Pellissier et al., 2023).
* Male and female.
* Normal BMI ranges between 18.5:24.9 kg/m2.

exclusion criteria:

* Physiotherapists outside the target range age an BMI.
* Students of physical therapy or Physiotherapists who worked for less than two years.
* Physiotherapists who had lumbar spine surgery.
* Physiotherapists who had history sever lumbar problem spondylolisthesis, tumor, fracture.
* Physiotherapists who suffers from vertigo.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-04 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
intensity of low back pain | 1 month
  we will assess intensity of low back pain by using visual analogue scale

SECONDARY OUTCOMES:
back muscle endurance | 1 month
  assess back muscle endurance by using Sorensen test
level of function (disability) associated with mechanical Low Back Pain | 1 month
  the Arabic version of Oswestry Disability Index will be used to determine the level of function associated with mechanical Low Back Pain
Fatigue Severity | 1 month
  The Arabic version of The Fatigue Severity Scale will be used to measure fatigue in people with mechanical Low Back Pain
psycho-social factors at work | 1 month
  The English version of The Brief Job Stress Questionnaire which is valid in the measurement of psycho-social factors at work and this Questionnaire can be one of the methodological tools to explore the mechanisms between job stress and several work-related disorders and can provide hints of intervention.

REFERENCES:
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Vieira ER, Svoboda S, Belniak A, Brunt D, Rose-St Prix C, Roberts L, da Costa BR. Work-related musculoskeletal disorders among physical therapists: an online survey. Disabil Rehabil. 2016;38(6):552-7. doi: 10.3109/09638288.2015.1049375. Epub 2015 May 26. PMID 26007284
- [Background] Areeudomwong P, Buttagat V. Comparison of Core Stabilisation Exercise and Proprioceptive Neuromuscular Facilitation Training on Pain-related and Neuromuscular Response Outcomes for Chronic Low Back Pain: A Randomised Controlled Trial. Malays J Med Sci. 2019 Nov;26(6):77-89. doi: 10.21315/mjms2019.26.6.8. Epub 2019 Dec 30. PMID 31908589